CLINICAL TRIAL: NCT05382650
Title: Multicenter Safety Evaluation of Human Rabies Immune Globulin 300 IU/mL in Children
Brief Title: Survey of Human Rabies Immune Globulin Safety in Children
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Principal Investigator, Michael Sirimaturos, Administrative Specialist - System Critical Care Services Leader, The Methodist Hospital Research Institute
Other Study IDs: PRO00028137
Record Dates: First submitted 2022-04-28; First posted 2022-05-19 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Rabies; Rabies Human; Rabies Virus Infection; Pediatrics
Keywords: Pediatrics; Rabies post-exposure prophylaxis; Rabies PEP; Rabies immune globulin; Rabies IG; Adverse events
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Biological: Human rabies immune globulin 300 IU/mL — All participants in this single-cohort observational study will receive human rabies immune globulin 300 IU/mL at a dose of 20 IU/kg per standard of care.

SUMMARY:
This observational study will be conducted across the Houston Methodist system, including all hospital-based and freestanding emergency departments (ED), and up to 4 additional sites in the United States. The safety of human rabies immune globulin (HRIG) 300 IU/mL product (HyperRAB®) in pediatric patients has not been fully established. The purpose of this study is to evaluate the safety of HRIG 300 IU/mL when given to pediatric patients per standard of care for rabies postexposure prophylaxis (PEP) in the ED.

DETAILED DESCRIPTION:
BACKGROUND: Rabies PEP consists of thorough wound cleansing, administration of HRIG 20 IU/kg body weight, and 4 to 5 doses of rabies vaccine. The safety of HRIG 300 IU/mL has been confirmed only for adult patients. Although the safety of HRIG 300 IU/mL in the pediatric population has not been fully established, there is no age limit on the FDA approved indication for HRIG 300 IU/mL, and it is routinely administered to pediatric patients as standard of care in the United States.

STUDY DESIGN: This observational, multicenter, prospective study will collect information on safety events that occur up to 30 days after standard of care administration of HRIG 300 IU/mL among pediatric patients (age ≤17 years) at up to 5 study sites in the United States. Safety data will be collected using surveys and chart review of the health record. All participants will receive HRIG 300 IU/mL per standard of care prior to joining this study. The day of HRIG 300 IU/mL administration will be defined as day 0. The study will conduct Survey 1 on day 2 and Survey 2 on day 10 to collect information on adverse events (AEs). Investigators will review the electronic health record on day 30 to collect additional information on AEs. If a serious adverse event is detected during Survey 1, Survey 2, or the 30-day chart review and is not previously documented as being resolved or stabilized the study will conduct Survey 3 on day 30.

ELIGIBILITY:
Inclusion Criteria

1. Received HRIG 300 IU/mL for rabies PEP during an ED encounter visit
2. Aged ≤17 years

Exclusion Criteria

1. HRIG 300 IU/mL dose given is <18 IU/kg or >22 IU/kg
2. Patient is admitted or transferred to a hospital from the ED for further management of injuries related to the animal exposure
3. Patient has a history of rabies vaccine or rabies immune globulin administration
4. Legally authorized representative (parent) does not speak English if patient is <7 years old
5. Legally authorized representative (parent) or patient does not speak English if patient is 7 to 17 years old
6. Inability to obtain consent

   1. More than 3 days passed since HRIG 300 IU/mL administration prior to screen
   2. Unable to contact legally authorized representative (parent) and/or patient within 3 days of HRIG 300 IU/mL administration
   3. Legally authorized representative (parent) and/or patient declined participation
7. Administration sites for HRIG are unknown

Max Age: 17 Years | Sex: All
Age Groups: Child
Study Population: Pediatric patients who received HRIG 300 IU/mL as part of routine medical care for rabies PEP during an ED visit in up to 5 study sites in the United States
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Incidence of local and systemic adverse events (AEs) within 2 days of HRIG 300 IU/mL administration | Within 2 days of HRIG 300 IU/mL administration
  Proportion of patients with 1 or more AEs deemed as possibly/definitely related to HRIG 300 IU/mL administration

SECONDARY OUTCOMES:
Cumulative incidence of all local and systemic AEs within 10 days of HRIG 300 IU/mL administration | Within 10 days of HRIG 300 IU/mL administration
  Proportion of patients with 1 or more AEs deemed as possibly/definitely related to HRIG 300 IU/mL administration
Cumulative incidence of all local and systemic AEs within 30 days of HRIG 300 IU/mL administration | Within 30 days of HRIG 300 IU/mL administration
  Proportion of patients with 1 or more AEs deemed as possibly/definitely related to HRIG 300 IU/mL administration
Cumulative incidence of all local and systemic serious adverse events (SAEs) within 30 days of HRIG 300 IU/mL administration | Within 30 days of HRIG 300 IU/mL administration
  Proportion of patients with 1 or more SAE deemed as possibly/definitely related to HRIG 300 IU/mL administration. An AE is considered "serious" if any of the following outcomes occur:
  * Death
  * Life-threatening AE (life-threatening in the definition of "serious" refers to an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)
  * In-patient hospitalization or prolongation of existing hospitalization
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * An important medical event (refers to events which may not be immediately life-threatening, or result in death, or hospitalization, but from medical and scientific judgment, may jeopardize the participant or/and may require medical or surgical intervention to prevent one of the other outcomes listed above).
Type and severity of individual local and systemic AEs detected within 30 days of HRIG 300 IU/mL administration | Within 30 days of HRIG 300 IU/mL administration
  Proportions of AEs that are local vs systemic and proportions of AEs that are mild, moderate, or severe among AEs deemed as possibly/definitely related to HRIG 300 IU/mL administration

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sirimaturos, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (2):
- United States (2):
  - Houston Methodist, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manning SE, Rupprecht CE, Fishbein D, Hanlon CA, Lumlertdacha B, Guerra M, Meltzer MI, Dhankhar P, Vaidya SA, Jenkins SR, Sun B, Hull HF; Advisory Committee on Immunization Practices Centers for Disease Control and Prevention (CDC). Human rabies prevention--United States, 2008: recommendations of the Advisory Committee on Immunization Practices. MMWR Recomm Rep. 2008 May 23;57(RR-3):1-28. PMID 18496505
- [Background] Hwang GS, Rizk E, Bui LN, Iso T, Sartain EI, Tran AT, Swan JT. Adherence to guideline recommendations for human rabies immune globulin patient selection, dosing, timing, and anatomical site of administration in rabies postexposure prophylaxis. Hum Vaccin Immunother. 2020;16(1):51-60. doi: 10.1080/21645515.2019.1632680. Epub 2019 Aug 1. PMID 31210569
- [Background] Hanna K, Cruz MC, Mondou E, Corsi E, Vandeberg P. Safety and neutralizing rabies antibody in healthy subjects given a single dose of rabies immune globulin caprylate/chromatography purified. Clin Pharmacol. 2018 Jun 26;10:79-88. doi: 10.2147/CPAA.S166454. eCollection 2018. PMID 29983597
- See also: Kamada Ltd., Kedrion Biopharma. U.S. Post-Marketing Pediatric Trial of a Human Rabies Immune Globulin (HRIG). Accessed April 11, 2022 — https://www.globenewswire.com/news-release/2020/08/19/2080546/0/en/Kamada-and-Kedrion-Biopharma-Announce-Results-of-First-and-Only-U-S-Post-Marketing-Pediatric-Trial-of-a-Human-Rabies-Immune-Globulin-HRIG-The-Study-Met-Its-Primary-Objective.html
- See also: Identifier NCT02912845, Post-marketing Study of KamRAB Administered as a Single Dose With Active Rabies Vaccine in Children Exposed to Rabies. National Library of Medicine (US); 2019. Accessed April 11, 2022 — https://ClinicalTrials.gov/show/NCT02912845
- See also: Centers for Disease Control and Prevention. Rabies in the United States: Protecting Public Health. Accessed November 11, 2025 — https://www.cdc.gov/rabies/php/protecting-public-health/index.html
- See also: World Health Organization. Rabies. Accessed April 11, 2022 — https://www.who.int/en/news-room/fact-sheets/detail/rabies
- See also: HyperRab® [rabies immune globulin (human)] [package insert]. Grifols Therapeutics Inc., Research Triangle Park, NC, USA. 2021. Accessed April 11, 2022 — https://www.hyperrab.com/documents/2533658/2533707/Prescribing+Information+HyperRAB+300.pdf/813095ad-a0b7-48fd-b3a8-c531d418e148?t=1617208717698